CLINICAL TRIAL: NCT01598246
Title: Prospective Observational Study on Factors Influencing Re-Intubation Following a Planned Extubation (RIPE) in a Pediatric Intensive Care Unit: Identifying Targets for a Quality Improvement Initiative
Brief Title: Study to Evaluate Causes of Failure to Extubate
Acronym: RIPE
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02-051E
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Extubation Failures
Keywords: Extubation failures; Sedation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extubation Success: Patients who do not require re-intubation, upto 72 hours after a planned extubation in the pediatric intensive care unit.
- Extubation failure: Patients who required re-intubation within 72 hours after a planned extubation in pediatric intensive care unit. To be further classified as early <12 hour and late 12-72 hour, extubation failures.

SUMMARY:
This is a prospective chart review of all extubations in the pediatric intensive care unit. Over a one year period all extubations in the unit are to be recorded on a designated form and standard variables charted and compared. All data will be collected from the chart, retrospectively after the extubation event. Patients who fail extubation will be compared to those who succeed. We aim to identify factors which contribute to extubation failures in the unit, to come up with a unit specific extubation policy

DETAILED DESCRIPTION:
Description of project- This is a prospective chart review to identify factors influencing a successful extubation event.

Hypothesis- Successful extubation in a pediatric intensive care unit is dependent on variables, which can be identified and the chances of success predicted. A clinical practice based upon such a prediction model, will improve the quality of care provided to the patients.

Type- Prospective chart review .

Procedure- Over 1 year period, all planned extubations in the intensive care unit to be recorded on a designated form and standard variables charted. All extubation decisions are to be made by the covering attending physician and at no time, the study protocol will affect/influence or alter the standard patient care. All data will be collected retrospectively after the extubation event. All included patients will be assigned a unique identification number (UID) by the investigator, who will secure the patient identifiers in an encrypted electronic file. Extubation failure will be defined as reintubation within 72 hours of a planned extubation and will be further classified as early (<12 hours) and late (12-72 hours) extubation failure. The cause of extubation failure will be recorded (as identified by the attending physician on service, who is not involved in the study).

Data collection and statistical analysis- The data will be collected on a standard form. The data collected will be periodically logged in an electronic data base and analyzed. Investigators will perform an interim analysis at the end of 6 months and a final analysis of the data at the end of 1 year period. Since this is an observational study, all the extubations in the time period, will be included. Based on 2010 data collected, for monitoring unplanned extubations (300 extubations) and considering recent expansion in their unit, investigators expect about 500 extubations in the time period.

For statistical analysis, group that fail extubation, will be compared, with the group that was an extubation success. Standard demographics (age, sex), patient disease related factors (diagnosis, duration of intubation, secretions, sedation level), care factors (CPAP trials, cuff leak test, use of pre-extubation decadron, p/f ratio prior to extubation), and post extubation care (post extubation respiratory support, stridor, blood gas) along with any complication during extubation and reintubation and reasons for reintubation will be collected and compared. As two groups are being compared, bivariate analyses utilizing Chi-square tests or univariate logistic regression for categorical variables and Student t -tests for interval variables, will be done. Based on 9.9% extubation failure rate in 2010, investigators expect ~50 extubation failures in the time frame. From the preliminary data, investigators also expect a 40% difference in the primary variables of comparison (age, secretions, sedation level). For statistical analysis at 95% confidence interval and 80% power, investigators will be able to detect differences between groups in proportions of approximately 20% with the expected sample size or differences of 25% with a 99% CI. The investigators also will conduct multivariate logistic regression analysis using extubation failure as the dependent variable and calculate the independent odds ratio for significant predictor variables. Early Vs late extubation failures, will also be compared. From literature, investigators assume 80% of extubation failures to be early (from their estimate, 40 early extubation failures and 10 late extubation failures, in 1 year period). They do not expect statistically significant results from the numbers in present trial period, however they expect to get trends to plan a further study.

ELIGIBILITY:
Inclusion Criteria:

* All planned extubations in pediatric Intensive care unit

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0 to 18 years, admitted in pediatric intensive care unit and required intubation and mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Tripathi, M.D, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical center, The Bronx, New York, United States